CLINICAL TRIAL: NCT06755489
Title: Evaluation of Quality of Life in a Cohort of Diarrhoeic Irritable Bowel Syndrome (IBS-D) Patients Assuming GABA.
Brief Title: Quality of Life in Diarrhea-predominant Irritable Bowel Syndrome Taking GABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Collaborators: Azienda Ospedaliero-Universitaria Pisana (AOUP) (Unknown)
Responsible Party: Principal Investigator, Massimo Bellini, Full professor in gastroenterology, University of Pisa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GABA 2.0
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diarrhoea Predominant Irritable Bowel Syndrome
Keywords: gamma-aminobutyric acid; diarrhoea; abdominal pain; irritable bowel syndrome; GABA
MeSH Terms: conditions — Diarrhea; Abdominal Pain; Irritable Bowel Syndrome | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, double-blind, parallel group, placebo-controlled, cross-over study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: Placebo; Other: GABA
- Group B (Experimental)
  Interventions: Other: Placebo; Other: GABA

INTERVENTIONS:
Other: Placebo — 530 mg tablets containing microcrystalline cellulose, rice bran, bitter cocoa powder table 530 mg. 1 tablet three times a day
Other: GABA — 530 mg tablets containing Gamma-aminobutyric acid (GABA) and different bulking agent as microcrystalline cellulose, calcium carbonate, lemon balm d.e. Leaves (melissa officinalis l. - maltodextrin) tit. 2% in rosmarinic acid, anti-caking agents: silicon dioxide, vegetable magnesium stearate. 1 tablet three times a day

SUMMARY:
The study aims to evaluate the impact on quality of life and abdominal discomfort of GABA and Melissa food supplement administration in patients with diarrhea-predominant irritable bowel syndrome.

DETAILED DESCRIPTION:
Rationale: Visceral pain represents a grievous form of pain that affects about 25% of the world population; abdominal pain is the most common gastrointestinal problem, encountered in a high percentage of adolescents, above all in women. It can be the result of prolonged inflammatory processes, such as in inflammatory bowel diseases (IBDs), but in many patients, negative diagnostic test results lead to the diagnosis of irritable bowel syndrome (IBS) .

Abdominal pain is a common manifestation in IBD, due to changes that begin with hypersensitivity of the primary sensory neurons, which innervate the gastrointestinal tract, and afterwards reach the central nervous system (CNS) . Inflammation does not seem to completely explain altered perception of pain in patients affect by IBD, as 20%-50% of patients complain about abdominal pain in the clinical remission stage . IBS is a functional bowel disorder characterized by the presence of chronic/recurrent abdominal pain or discomfort, with altered bowel habits and consequent anomalies in stool frequency and form . Pathogenesis of IBS is only partially understood, even though there is some evidence that changes in the digestive motility and secretion, visceral hypersensitivity, abnormalities of enteroendocrine and immune systems, genetic factors, infections, alterations of the intestinal microbiota and inflammation could play a role in this functional disease. . Patients may be categorized as diarrheal-predominant (IBS-D), constipation-predominant IBS-C), or as having both (IBS-M) . In this context, finding valid therapies that can alleviate chronic visceral pain represents an important medical need to improve patients' quality of life. Unfortunately, the current therapeutics to treat visceral pain offer little benefit for abdominal symptoms and can produce undesired and serious side effects . In this regard, the pain management remains unsatisfactory, so there is a growing demand for the development of effective treatments. Considering that visceral pain has been related to inflammatory processes , as well as to alterations in the enteric barrier and immune response , a product able to protect the intestinal mucosa by indirectly controlling inflammation and at the same time modulating immune response could be the answer. In this regard, gamma aminobutyric acid (GABA) is known to exert a number of beneficial effects at digestive level. For instance, GABA has a protective role during inflammatory processes by modulating cytokine production . Moreover, products containing GABA have been proven to strengthen intestinal epithelial barrier and to modulate immune-inflammatory response .

Objectives: Primary: to evaluate the changes in quality of life in IBS-D patients taking GABA food supplement. Secondary: evaluation of changes in abdominal discomfort in IBS-D patients taking GABA food supplement; evaluation of global symptom score in IBS-D patients taking GABA food supplement; self evaluation of psychological impact of IBS-D in patients taking GABA food supplement; intestinal microbiota changes in IBS-D patients taking GABA food supplement; evaluation of epithelial barrier impairment in IBS-D patients taking GABA food supplement; evaluation of systemic inflammation in IBS-D patients taking GABA food supplement.

Investigational product, dose, and mode of administration: Regimen A: EIRENE® (containing GABA and Melissa officials) food supplement table 530 mg, 1 tablet three times a day. Regimen B: placebo (microcrystalline cellulose, rice bran, bitter cocoa powder) table 530 mg, 1 tablet three times a day.

Methodology: This is a monocentric, randomized, double-blind, parallel group, placebo-controlled, 2-period cross-over study investigating the changes in quality of life, abdominal symptoms, intestinal microbiota, intestinal permeability, systemic inflammation in patients taking a GABA-based food supplement. Patients will be evaluated before and after each treatment period (Regimen A and Regimen B) through clinical questionnaires and scales, blood and stool tests.

The following questionnaires will be administered:

* Short-Form 36
* 11 points visual analogue scale for abdominal discomfort
* Hospital Anxiety and Depression Scale
* Bristol Stool Scale

The following evaluations will be performed on blood samples:

* TNF-alfa, IL-1β, C-reactive protein and IL-10 levels to assess systemic inflammation
* Lypopolisaccharide binding protein (LBP) to assess intestinal epithelial barrier impairment.
* Blood tests for safety (glucose, BUN, AST, ALT, bilirubin, ALP, creatinin, blood count and formula, platelets, Na, K, Ca)

The following evaluations will be performed on stool samples:

* Fecal calprotectin
* Fecal microbiome analysis

Inclusion criteria: Age > 18 years and ≤ 75; a positive diagnosis of IBS-D according to Rome IV criteria; both males and females; negative relevant additional screening or consultation whenever appropriate; colonoscopy if there are alarm symptoms (eg. Rectal bleeding, pseudodiarrhea. If the patients' age is > or = 50 yrs a colonoscopy within 5 years is mandatory); availability to participate in the clinical study, confirmed by the signed informed consent form; ability to conform to the study protocol; patients' ability to complain study protocol procedures; subjects who decide to use single or double contraceptive methods not to conceive during study period.

Exclusion criteria: patients with IBS-C, IBS-M and IBS-U according to Rome IV criteria; presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant; ascertained intestinal organic diseases, including celiac disease, food allergies or inflammatory bowel diseases (Crohn's disease, ulcerative colitis, diverticular disease, infectious colitis, ischemic colitis, microscopic colitis); previous major abdominal surgery; active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrollment are also acceptable); use of -pre or probiotics, topical and/or systemic antibiotic and prokinetic therapy during the 15 days before treatment starts; systematic/frequent use of contact laxatives; pregnant or breastfeeding woman; females of childbearing potential in the absence of effective contraceptive methods; inability to conform to protocol; treatment with any investigational drug within the previous 30 days; recent history or suspicion of alcohol abuse or drug addiction; presence of red or white flags at the Rome IV Psychosocial Alarm Questionnaire for Functional gastrointestinal Disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and ≤ 75
* A positive diagnosis of IBS-D according to Rome IV criteria.
* Both males and females.
* Negative relevant additional screening or consultation whenever appropriate
* Colonoscopy if there are alarm symptoms (eg. Rectal bleeding, pseudodiarrhea). If the patients' age is > or = 50 yrs a colonoscopy within 5 years is mandatory.
* Availability to participate in the clinical study, confirmed by the signed informed consent form.
* Ability to conform to the study protocol.
* Patients' ability to complain study protocol procedures.
* Subjects who decide to use single or double contraceptive methods not to conceive during study period.

Exclusion Criteria:

* Patients with IBS-C, IBS-M and IBS-U according to Rome IV criteria.
* Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant.
* Ascertained intestinal organic diseases, including celiac disease, food allergies or inflammatory bowel diseases (Crohn's disease, ulcerative colitis, diverticular disease, infectious colitis, ischemic colitis, microscopic colitis).
* Previous major abdominal surgery.
* Active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment are also acceptable).
* Use of -pre or probiotics, topical and/or systemic antibiotic and prokinetic therapy during the 15 days before treatment starts.
* Systematic/frequent use of contact laxatives.
* Pregnant or breastfeeding woman.
* Females of childbearing potential in the absence of effective contraceptive methods.
* Inability to conform to protocol.
* Treatment with any investigational drug within the previous 30 days.
* Recent history or suspicion of alcohol abuse or drug addiction.
* Presence of red or white flags at the Rome IV Psychosocial Alarm Questionnaire for Functional gastrointestinal Disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Quality of life | From enrollment to the end of treatment at 12 weeks. Evaluated at every scheduled visit (V0, V1, V2, V3, FU)
  Evaluation of quality of life in IBS-D patients taking GABA food supplement with Short-Form 36 Items Health Survey (SF-36 Italian version). A reduction at least of 10 points on at least 1 of the 8 subdomains of the SF36 score would be considered significant.

SECONDARY OUTCOMES:
Abdominal discomfort | From enrollment to the end of treatment at 12 weeks. Evaluated at every scheduled visit (V0 (Week0), V1(Week 4), V2(Week 6), V3(week 10), FU(Week 12))
  Abdominal discomfort evaluated by a 11 points visual analogue scale
Psychological impact | From enrollment to the end of treatment at 12 weeks. Evaluated at every scheduled visit (V0, V1, V2, V3, FU)
  Self evaluation of psychological impact of IBS-D in patients taking GABA food supplement with Hospital Anxiety and Depression Scale (HADS).
Intestinal microbiota | From enrollment to the end of treatment at 10 weeks. Evaluated at every scheduled visit (V0, V1, V2, V3)
  Microbiota changes in IBS-D patients taking GABA food supplement with NGS analysis. Results will be evaluated describing variations of principal genera and family variation.
Epithelial barrier impairment | From enrollment to the end of treatment at 10 weeks. Evaluated at every scheduled visit (V0, V1, V2, V3)
  Evaluation of epithelial barrier impairment in IBS-D patients taking GABA food supplement with haematological dosage of Lypopolisaccharide binding protein (LBP).
Systemic inflammation | From enrollment to the end of treatment at 10 weeks. Evaluated at every scheduled visit (V0, V1, V2, V3)
  Evaluation of systemic inflammation in IBS-D patients taking GABA food supplement with haematological dosage of TNF-alfa, IL-1β, C-reactive protein and IL-10 levels

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - University of Pisa, Pisa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Sokovic Bajic S, Djokic J, Dinic M, Veljovic K, Golic N, Mihajlovic S, Tolinacki M. GABA-Producing Natural Dairy Isolate From Artisanal Zlatar Cheese Attenuates Gut Inflammation and Strengthens Gut Epithelial Barrier in vitro. Front Microbiol. 2019 Mar 18;10:527. doi: 10.3389/fmicb.2019.00527. eCollection 2019. PMID 30936860
- [Background] Gros M, Gros B, Mesonero JE, Latorre E. Neurotransmitter Dysfunction in Irritable Bowel Syndrome: Emerging Approaches for Management. J Clin Med. 2021 Jul 31;10(15):3429. doi: 10.3390/jcm10153429. PMID 34362210
- [Background] Carabotti M, Scirocco A, Maselli MA, Severi C. The gut-brain axis: interactions between enteric microbiota, central and enteric nervous systems. Ann Gastroenterol. 2015 Apr-Jun;28(2):203-209. PMID 25830558
- [Background] Cervero F. Central sensitization and visceral hypersensitivity: Facts and fictions. Scand J Pain. 2014 Apr 1;5(2):49-50. doi: 10.1016/j.sjpain.2014.02.005. No abstract available. PMID 29913675
- [Background] Bellini M, Gambaccini D, Stasi C, Urbano MT, Marchi S, Usai-Satta P. Irritable bowel syndrome: a disease still searching for pathogenesis, diagnosis and therapy. World J Gastroenterol. 2014 Jul 21;20(27):8807-20. doi: 10.3748/wjg.v20.i27.8807. PMID 25083055
- [Background] Portincasa P, Bonfrate L, de Bari O, Lembo A, Ballou S. Irritable bowel syndrome and diet. Gastroenterol Rep (Oxf). 2017 Feb;5(1):11-19. doi: 10.1093/gastro/gow047. Epub 2017 Jan 20. PMID 28110300
- [Background] Minderhoud IM, Oldenburg B, Wismeijer JA, van Berge Henegouwen GP, Smout AJ. IBS-like symptoms in patients with inflammatory bowel disease in remission; relationships with quality of life and coping behavior. Dig Dis Sci. 2004 Mar;49(3):469-74. doi: 10.1023/b:ddas.0000020506.84248.f9. PMID 15139501
- [Background] Morales-Soto W, Gulbransen BD. Enteric Glia: A New Player in Abdominal Pain. Cell Mol Gastroenterol Hepatol. 2019;7(2):433-445. doi: 10.1016/j.jcmgh.2018.11.005. Epub 2018 Nov 24. PMID 30739868